CLINICAL TRIAL: NCT06780397
Title: Monocentric Study on the Clinical and Ultrasound Incidence of Rheumathologic Immune Related Adverse Events in Patients Affected by Stage IIB, IIC, III and IV Melanoma Under Therapy With Immune-checkpoint Inhibitors
Brief Title: Clinical and Ultrasound Incidence of Rheumatologic Immune Related Adverse Events in Stage IIB-IV Melanoma Patients
Acronym: Mel-Immuno-Reu
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6839
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Melanoma, Stage II; Melanoma Stage III; Melanoma Stage IV
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Joint ultrasonography — Patients will undergo rheumatologic visits at baseline and scheduled follow-ups.
  Rheumatologic visit procedures:
  * collection of patients' anamnesis of rheumatologic diaseases.
  * identification of painful and/or swollen joints and enthesis.
  * evaluation of joint and enthesis pain.
  * joint ultrasonography and assessment of joint structures and enthesis.
Other: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 version 3.0 — Patients will undergo dermatologic visits at baseline and scheduled follow-ups.
  Dermatologic visit procedures:
  * collection of patients' oncologic anamnesis and general personal and lifestyle information.
  * administration of the quality of life questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 version 3.0) to assess the impact of rheumatologic adverse events on patients' quality of life.

SUMMARY:
Rheumatologic adverse events are expected to affect between 3% and 7.5% of patients undergoing immunotherapy and are likely to be underdiagnosed.

The main aim of this observational prospective study is to investigate the clinical and ultrasonographic incidence of rheumathologic immune related adverse events in a cohort of patients affected by stage IIB, IIC, III and IV melanoma undergoing treatment with immune-checkpoint inhibitors.

Patients will:

* receive immune-checkpoint inhibitor therapy, according to disease stage and current National Guidelines.
* undergo dermatologic visit prior to the start of immune-checkpoint inhibitor therapy and at scheduled follow-ups.
* undergo rheumatologic visit prior to the start of immune-checkpoint inhibitor therapy and at scheduled follow-ups.
* receive a quality of life questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 version 3.0) prior to the start of immune-checkpoint inhibitor therapy and at scheduled follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients affected by stage IIB, IIC, III and IV melanoma who start systemic therapy with immune-checkpoint inhibitors.
* Signature of the patient consent to the study.

Exclusion Criteria:

* Patients aged below 18 years of age.
* Patients who are unable to express consent to the study.
* Patients with a diagnosis of chronic joint diseases: inflammatory arthritis, arthrosis, microcrystalline arthritis, septic arthritis etc.
* Systemic diseases with likely joint involvement (inflammatory bowel disease, etc.)
* Previous treatments with immune-checkpoint inhibitors or previous adjuvant therapy with immune-checkpoint inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients affected by stage IIB-IV melanoma who start systemic therapy with immune-checkpoint inhibitors.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Investigation of the incidence of rheumatologic immune related adverse events during immune-checkpoint inhibitor treatment in stage IIB-IV melanoma patients. | 3 years
  Patients will undergo a rheumatologic visit and joint ultrasonography at baseline and at scheduled follow-ups in order to assess the incidence of rheumatologic immune related adverse events.

SECONDARY OUTCOMES:
Description of the main characteristics of the rheumatologic immune related adverse events in stage IIB-IV melanoma patients under immune-checkpoint inhibitor therapy. | 3 years
  A rheumatologist will clinically and ultrasonographically characterize the main features of the rheumatologic immune related adverse events occuring during immunotherapy.
Identification of baseline risk factors associated with occurrence of rheumatologic immune related adverse events in stage IIB-IV melanoma patients under immune-checkpoint inhibitor therapy. | 3 years
  Baseline clinical, dermatological, rheumatologic and ultrasonographic factors will be recorded and associated with the occurrence of rheumatologic immune related adverse events during immunotherapy.
Evaluation of rheumatologic adverse events impact on patients' quality of life. | 3 years
  Patients will receive a quality of life questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 version 3.0) at baseline and at scheduled timepoints, in order to investigate the impact of the occurrence of rheumatologic adverse events on patients' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ketty Peris, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Dermatologia, Rome, Lazio, Italy